CLINICAL TRIAL: NCT07316322
Title: Comparison of Central Sensitization in Painful and Painless Diabetic Peripheral Neuropathy Phenotypes: A Multidimensional Psychophysiological Assessment
Brief Title: Central Sensitization in Painful and Painless Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Doctor Lecturer, Inonu University
Other Study IDs: 1003
Record Dates: First submitted 2025-12-15; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus (DM)
Keywords: Diabetus Mellitus; Central sensitization; Temporal summation; Neuropathic pain
MeSH Terms: conditions — Diabetes Mellitus; Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Painful DPN Group: The study will include individuals aged 18-80 years who have been diagnosed with diabetic neuropathy, show a positive result on the MNSI-clinical assessment, and have a DN4 score of ≥4.This study is entirely observational and cross-sectional in nature, and no therapeutic intervention will be administered to the participants.
- Painless DPN Group: The study will include individuals aged 18-80 years who have been diagnosed with diabetes mellitus, have a positive MNSI-clinical assessment, and a DN4 score of <4. This study is entirely observational and cross-sectional in nature, and no therapeutic intervention will be administered to the participants.
- Diabetic Control Group Without Diabetic Peripheral Neuropathy (DPN): The study will include individuals aged 18-80 years who have been diagnosed with diabetes mellitus, have a negative MNSI-clinical assessment, and a DN4 score of <4. This study is entirely observational and cross-sectional in nature, and no therapeutic intervention will be administered to the participants.
- Healthy Control Group: The study will include individuals aged 18-80 years who do not have a diagnosis of diabetes mellitus, have a negative MNSI-clinical assessment, and a DN4 score of <4. This study is entirely observational and cross-sectional in nature, and no therapeutic intervention will be administered to the participants.

SUMMARY:
This research is structured as a cross-sectional observational study. The primary objective is to compare central sensitization across painful and painless phenotypes of diabetic peripheral neuropathy. The study will be conducted among individuals diagnosed with type 2 diabetes mellitus at the Department of Geriatrics, İnönü University Turgut Özal Medical Center. All assessments will be administered in accordance with a rigorously standardized protocol.

Eligible participants will include individuals aged 18 to 80 years who have had a confirmed diagnosis of type 2 diabetes mellitus for at least one year, are capable of comprehending and following verbal instructions in Turkish required for the study procedures, and provide written informed consent.

All statistical analyses will be performed using IBM SPSS Statistics (v.29, Armonk, NY, USA) and JASP (v.0.18, Amsterdam, Netherlands).

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a well-known metabolic disease characterized by organ dysfunction that arises directly or indirectly from the effects of chronic hyperglycemia, affecting a substantial portion of the global population. According to the International Diabetes Federation, the global prevalence of diabetes was estimated at 9.3% in 2019, with 463 million individuals living with the disease, and this prevalence is projected to rise to 10.2% (578 million) by 2030 and 10.9% (700 million) by 2045. Both Type 2 Diabetes (T2DM) and Type 1 Diabetes (T1DM) lead to elevated glucose concentrations and increased inflammatory processes, resulting in a wide range of complications including diabetic retinopathy, diabetic nephropathy, diabetic neuropathy, cardiovascular diseases, musculoskeletal disorders, impaired fracture and wound healing, and pain. Diabetic polyneuropathy (DPN) is a clinical syndrome characterized by pain associated with lesions of the somatosensory nervous system. Between 10-20% of individuals with diabetes experience pain due to the presence of peripheral neuropathy, and there is no universally accepted gold standard for diagnosing DPN; accurately identifying painful DPN remains challenging, particularly because neuropathic pain is often difficult to distinguish from non-neuropathic pain. The mechanisms of neuropathic pain are complex. Peripheral tissue damage can trigger peripheral sensitization; however, central sensitization of the central nervous system plays the predominant role. DM may affect central nervous system processes, leading to central sensitization and dysfunction of pain modulation. Central sensitization is defined as an increased responsiveness of the central nociceptive system, which contributes to the amplification and spread of pain. Recent studies over the past five years have demonstrated that central neuropathic mechanisms may contribute to diabetes-related pain, similar to other neuropathic pain conditions. While there is extensive literature evaluating diabetic neuropathic pain, studies specifically investigating nociceptive pain remain limited. The primary aim of this study is to compare central sensitization across painful and painless diabetic peripheral neuropathy phenotypes.This research is planned as a cross-sectional observational study. It will be conducted in individuals diagnosed with Type 2 diabetes at the Department of Geriatrics, Turgut Özal Medical Center, İnönü University. All assessments will be performed according to a predetermined standardized protocol. Individuals aged 18-80 years who have had a diagnosis of Type 2 diabetes mellitus for at least one year and who can understand and follow verbal instructions in Turkish will be included. Initially, data regarding age, height, weight, smoking and alcohol use, duration of diagnosis, comorbidities, current medications and duration of use, biochemical test results, surgical history, and educational and income levels will be collected. Body mass index will be calculated for all participants. All statistical analyses will be conducted using IBM SPSS Statistics (v.29, Armonk, NY, USA) and JASP (v.0.18, Amsterdam, Netherlands). Descriptive data will be presented as mean ± SD for continuous variables and as percentages/frequencies for categorical variables. Data distribution will be assessed using the Shapiro-Wilk test. Between-group comparisons for continuous variables will be performed using one-way ANOVA or the Kruskal-Wallis test depending on distribution; when significant differences are identified, Tukey HSD or Dunn-Bonferroni post-hoc analyses will be conducted. Categorical variables will be analyzed using chi-square or Fisher's exact tests. Between-group differences will be further examined using one-way ANCOVA, with age, sex, HbA1c, diabetes duration, BMI, MNSI-clinical score, and DN4 score included as covariates. Effect sizes will be reported as partial eta-squared (η²ₚ) for interaction effects and Cohen's d for pairwise comparisons. Correlation analyses will be performed using Pearson or Spearman methods. Effect size assumptions were based on findings from a previous study investigating CPM effectiveness in individuals with diabetic polyneuropathy. That study reported mean CPM values of approximately -7.4 ± 1.0 in the painful DPN group and -2.3 ± 1.6 in the painless DPN group, yielding a mean difference of 5.1 and a pooled SD of 1.35, corresponding to Cohen's d ≈ 0.6. When adapted to a three-group phenotypic design, this effect size was converted to f ≈ 0.30 using the formula f = d / 2. Using these parameters (f = 0.30, α = 0.05, power = 0.80, number of groups = 3), a priori power analysis yielded a required sample size of 111 participants. Accounting for potential data loss, the sample size was increased by 15%, resulting in a final target of 128 participants (approximately 42-43 per group).

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 80 years of age
* Having a diagnosis of Type 2 diabetes mellitus for at least 1 year
* Providing written informed consent to participate in the study

Exclusion Criteria:

* Non-diabetic causes of polyneuropathy (alcohol, chemotherapy, vitamin deficiencies, renal failure, hypothyroidism, etc.)
* Active ulcer, infection, or severe vascular insufficiency in the lower extremity
* Central nervous system disorders (stroke, multiple sclerosis, spinal cord injury, etc.)
* Skin lesions, dermatitis, wounds, or infection in the test areas (foot or forearm)
* Peripheral entrapment neuropathies or related radiculopathies (e.g., carpal tunnel syndrome, C7-C8 radiculopathy)
* Chronic widespread pain syndrome (fibromyalgia, etc.) or active flaring rheumatologic disease
* Dose change within the last 2-4 weeks in medications affecting pain modulation (gabapentinoids, SNRI/TCA, opioids, hypnotics, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-80 who have had a diagnosis of Type 2 diabetes for at least 1 year will be included in this study.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Conditioned Pain Modulation (CPM) Test | Immediately before cuff inflation and immidiately after completion of the conditioning protocol
  Assessment will be performed using an algometer. The algometer probe is positioned perpendicularly over the trapezius muscle. Pressure is increased at a rate of approximately 30 kPa/s. When the participant first perceives pain, the measurement is stopped and this value is recorded as PPT₁ (pre-test). Conditioning Stimulus (CS) - To evaluate ischemic pain, a blood pressure cuff is placed on the participant's non-dominant arm and rapidly inflated to 240 mmHg. The participant is then instructed to perform repeated hand-opening and closing exercises involving the distal arm (forearm muscles) for approximately 2 minutes. When the participant reports pain intensity as NRS ≥ 7/10, the conditioning stimulus is considered adequate. For the repeated PPT measurement, while the cuff remains inflated, PPT is measured again at the same location. This value is recorded as PPT₂ (post-test). The CPM effect is calculated using the formula: CPM effect = PPT₂ - PPT₁.

SECONDARY OUTCOMES:
Central Sensitization Inventory (CSI) | Baseline(First assesstment
  The Central Sensitization Inventory (CSI) is a recently developed self-report screening tool designed to help identify patients with Central Sensitization Syndromes, including fibromyalgia. It consists of 25 items, each scored on a scale from 0 to 4, yielding a total score ranging from 0 to 100. Scores of 50 or higher indicate a very high level of central sensitization.
DN4 (Douleur Neuropathique) | Baseline(First assesstment)
  The DN4 (Douleur Neuropathique) questionnaire consists of sensory symptoms reported by the patient (7 items) and findings evaluated during physical examination (3 items). Each 'yes' response is scored as 1 point and each 'no' response as 0 points. The total score ranges from 0 to 10. A score of 4 or higher is considered indicative of neuropathic pain.
Michigan Neuropathy Screening Instrument (MNSI) | Baseline(First assesstment)
  The Michigan Neuropathy Screening Instrument (MNSI) is a two-part scale used to assess diabetic neuropathy. The first part consists of questions completed by the patient, while the second part is based on the clinician's physical examination. Some items are scored as 'yes = 1 point, no = 0 points,' whereas the opposite scoring applies to certain other items. The maximum total score is 13, and scores of 7 or higher indicate a significant risk of symptomatic neuropathy.
Numerical Rating Scale (NRS) | Baseline(First assesstment)
  Pain intensity will be assessed using the Numerical Rating Scale (NRS). The NRS is a unidimensional measure of pain severity primarily used in adults. Several versions exist, but the 11-point format is the most widely utilized. Using the NRS, patients report a number between 0 and 10 that best represents their pain intensity, where 0 indicates no pain and 10 represents the worst imaginable pain experienced within the past 24 hours.
Pain Catastrophizing Scale | Baseline(First assesstment)
  The Pain Catastrophizing Scale is a self-report questionnaire developed to measure the extent to which individuals catastrophize in response to pain. The 13-item scale, scored on a five-point Likert format, consists of three subcomponents: rumination, magnification, and helplessness. The rumination subscale score is calculated using responses to items 8, 9, 10, and 11. Each item is scored from 0 to 4, and the total score is obtained by summing all 13 items, yielding a range of 0-52. Scores of 30 or higher indicate high levels of catastrophizing, reflecting an increased risk of pain chronification.
Tampa Scale of Kinesiophobia | Baseline(First assesstment)
  The Tampa Scale of Kinesiophobia is a 17-item instrument developed to assess fear of movement and reinjury. The scale includes parameters related to work-associated activities, fear of injury/reinjury, and fear-avoidance beliefs. Each item is scored from 1 to 4, yielding a minimum score of 17 and a maximum score of 68. Scores of 37 or higher indicate a high level of kinesiophobia.
Hospital Anxiety and Depression Scale (HADS) | Baseline(First assesstment)
  The Hospital Anxiety and Depression Scale (HADS) consists of two subscales assessing anxiety and depression. It is a self-report instrument comprising 14 items, with 7 items evaluating depression (even-numbered items) and 7 items assessing anxiety (odd-numbered items). Responses are rated on a four-point Likert scale and scored from 0 to 3, with a maximum score of 21 for each subscale. Scores of 11 or higher indicate clinically significant levels of anxiety or depression. The purpose of the scale is not to establish a diagnosis but to rapidly screen for anxiety and depression in individuals with physical illness and identify those at risk.
Pittsburgh Sleep Quality Index (PSQI) | Baseline(First assesstment)
  The Pittsburgh Sleep Quality Index (PSQI) consists of 24 items in total. It includes seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. Higher total scores indicate poorer sleep quality. A global PSQI score of 5 or higher is considered indicative of poor sleep quality.
Temporal Summation | Baseline(First assesstment)
  Temporal summation will be assessed using a Semmes-Weinstein 26 g (~256 mN) monofilament. The participant is seated in a comfortable, supported position. Pain intensity is rated using the NRS. The monofilament is applied perpendicularly to the skin and bent to its buckling point within 1 second. Pain following the initial stimulus is recorded as NRS₁. Ten consecutive stimuli are then applied at the same site at a frequency of 1 Hz (using a metronome). Pain immediately after the 10th stimulus is recorded as NRS₂. Two trials are performed at each site (T1 → S10), with ≥60 seconds between trials. The mean of the two trials is used for analysis. The same procedure is repeated at the second site in a randomized order. Test Sites: Dorsum of the foot (dominant side; between the II-III metatarsal heads), distal/peripheral site, Dorsum of the forearm (dominant side; distal one-third of the radial dorsum) non-neuropathic control site.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynal Yasacı, Principal Investigator — Inonu University
Locations (1):
- Inonu University Turgut Ozal Medical Center, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data will be securely stored by the investigators and may be shared with authorized personnel if deemed necessary, in accordance with applicable privacy regulations.

REFERENCES:
- [Background] Granovsky Y, Shafran Topaz L, Laycock H, Zubiedat R, Crystal S, Buxbaum C, Bosak N, Hadad R, Domany E, Khamaisi M, Sprecher E, Bennett DL, Rice A, Yarnitsky D. Conditioned pain modulation is more efficient in patients with painful diabetic polyneuropathy than those with nonpainful diabetic polyneuropathy. Pain. 2022 May 1;163(5):827-833. doi: 10.1097/j.pain.0000000000002434. PMID 34371518
- [Background] İrem Mıhçıoğlu CM, Hacer Hicran Mutlu. Uykusuzluk Şikayetleri ve Uyku Kalitesi Temel Ölçeğinin Türkçe Geçerlilik ve Güvenirliği. 2017.
- [Background] Rabia Hacıhasanoğlu PK, Arzu Yıldırım,Seval Uslu, . Bir Sağlık Ocağına Başvuran Kronik Hastalığı Olan Bireylerde Anksiyete ve Depresyon 2010.
- [Background] Öznur Tunca Yılmaz YY, Fatma Uygur, Naime Uluğ Tampa Kinezyofobi Ölçeği'nin Türkçe versiyonu ve test-tekrar test güvenirliği 2011.
- [Background] Damla Karabay FT, Merve Keskin, Orhan Öztürk,Merve Kurt,Derya Özer Kaya. Ruminasyonun Tanınması ve Ağrı Deneyimi ve Fiziksel Aktivite ile İlişkisinin İncelenmesi: Geleneksel Derleme. 2023.
- [Background] Robinson CL, Phung A, Dominguez M, Remotti E, Ricciardelli R, Momah DU, Wahab S, Kim RS, Norman M, Zhang E, Hasoon J, Orhurh V, Viswanath O, Yazdi C, Chen GH, Simopoulos TT, Gill J. Pain Scales: What Are They and What Do They Mean. Curr Pain Headache Rep. 2024 Jan;28(1):11-25. doi: 10.1007/s11916-023-01195-2. Epub 2023 Dec 7. PMID 38060102
- [Background] Aktar Reyhanioglu D, Adiyaman SC, Bektas M, Bulut O, Ozgen Saydam B, Bayraktar F, Kara B. Validity and reliability of the Turkish version of the Michigan Neuropathy Screening Instrument. Turk J Med Sci. 2020 Jun 23;50(4):789-797. doi: 10.3906/sag-1906-63. PMID 32178509
- [Background] Unal-Cevik I, Sarioglu-Ay S, Evcik D. A comparison of the DN4 and LANSS questionnaires in the assessment of neuropathic pain: validity and reliability of the Turkish version of DN4. J Pain. 2010 Nov;11(11):1129-35. doi: 10.1016/j.jpain.2010.02.003. Epub 2010 Apr 24. PMID 20418179
- [Background] Düzce E. Santral Sensitizasyon Ölçeğinin Türkçe Geçerlilik ve Güvenilirliği. 2017.
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Fischer TZ, Waxman SG. Neuropathic pain in diabetes--evidence for a central mechanism. Nat Rev Neurol. 2010 Aug;6(8):462-6. doi: 10.1038/nrneurol.2010.90. Epub 2010 Jul 13. PMID 20625378
- [Background] Ma YC, Kang ZB, Shi YQ, Ji WY, Zhou WM, Nan W. The Complexity of Neuropathic Pain and Central Sensitization: Exploring Mechanisms and Therapeutic Prospects. J Integr Neurosci. 2024 Apr 25;23(5):89. doi: 10.31083/j.jin2305089. PMID 38812380
- [Background] Celik S, Yenidunya G, Temel E, Purisa S, Uzum AK, Gul N, Cinkil G, Dinccag N, Satman I. Utility of DN4 questionnaire in assessment of neuropathic pain and its clinical correlations in Turkish patients with diabetes mellitus. Prim Care Diabetes. 2016 Aug;10(4):259-64. doi: 10.1016/j.pcd.2015.11.005. Epub 2015 Dec 31. PMID 26749091
- [Background] Eitner A. [Diabetes mellitus-a risk factor for pain]. Schmerz. 2025 Oct;39(5):350-358. doi: 10.1007/s00482-025-00900-x. Epub 2025 Aug 28. German. PMID 40875021
- [Background] Lu Y, Wang W, Liu J, Xie M, Liu Q, Li S. Vascular complications of diabetes: A narrative review. Medicine (Baltimore). 2023 Oct 6;102(40):e35285. doi: 10.1097/MD.0000000000035285. PMID 37800828